CLINICAL TRIAL: NCT00980395
Title: A Phase II, Open-Label Study of Bortezomib (Velcade), Cladribine and Rituximab (VCR) in Advanced, Newly Diagnosed and Relapsed/Refractory Mantle Cell and Indolent Lymphomas
Brief Title: Bortezomib, Cladribine, and Rituximab in Treating Patients With Advanced Mantle Cell Lymphoma or Indolent Lymphoma
Acronym: VCR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0800001071; P30CA023074 (NIH); UARIZ-08-1071-04 (Other: UofA IRB); X05260 (Other: Sponsor Protocol ID); CDR0000655078 (Other: OLD PDQ #); 0800001071 (Other: UofA IRB #); 08-1071-04 (Other: UofA IRB #)
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Lymphoma; Mantle Cell Lymphoma; Indolent Lymphoma; SLL
Keywords: recurrent mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; Waldenstrom macroglobulinemia; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; extranodal marginal zone BCL mucosa assoc lymphoid tissue; nodal marginal zone B Cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — Rituximab; Bortezomib; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VCR (Velcade, Cladribine and Rituximab) (Experimental): * Rituximab 375 mg/m2 IV day1
  * Cladribine 4 mg/m2 IV over 2 hours days 1-5
  * Bortezomib 1.3 mg/m2 IV days 1 and 4
  * Repeat every 28 days for a maximum of 6 cycles
  Interventions: Drug: rituximab; Drug: bortezomib; Drug: cladribine

INTERVENTIONS:
Drug: rituximab — 375 mg/m2 IV Day 1. Repeat every 28 days for a maximum of 6 cycles.
  Other Names: Rituxan
Drug: bortezomib — 1.3 mg/m2 IV Days 1 and 4. Repeat every 28 days for a maximum of 6 cycles.
  Other Names: Velcade
Drug: cladribine — 4 mg/m2 IV over 2 hours Days 1-5. Repeat every 28 days for a maximum of 6 cycles.
  Other Names: Leustatin

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cladribine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with cladribine and rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with cladribine and rituximab works in treating patients with advanced mantle cell lymphoma or indolent lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 2-year progression-free survival of patients with advanced mantle cell lymphoma or indolent lymphoma treated with bortezomib, cladribine, and rituximab.

Secondary

* Determine the 2-year overall survival of patients treated with this regimen.
* Determine the complete response and overall response rate in patients treated with this regimen.
* Describe the long- and short-term toxicity of this regimen in these patients.
* Determine the prognostic importance of Aurora kinase A in patients treated with this regimen.
* Determine the cytokine profiles for each lymphoma subtype and how they change with this regimen.
* Evaluate the prognostic importance of major carcinogenic pathways using tissue microarray.

OUTLINE: Patients receive bortezomib IV on days 1 and 4, cladribine IV over 2 hours on days 1-5, and rituximab IV on day 1. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and after course 1 for cytokine profile studies. Previously collected tissue samples are obtained for analysis of Aurora kinase A and B, Ki-67, cyclin D, Bcl-2, phosphor-HisH3, c-Met, and VEGF expression by using tissue microarray (IHC staining), reverse transcriptase-PCR, and/or western blotting.

After completion of study therapy, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary consent before performance of any study-related procedure
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Biopsy-proven mantle cell, marginal zone, lymphoplasmacytic, small lymphocytic lymphoma, or follicular lymphoma
* CD20-positive disease
* Patients with marginal zone, lymphoplasmacytic, small lymphocytic, or follicular lymphoma - at least one criterion for initiation of treatment must be met:

  * Symptomatic disease
  * Cytopenia related to lymphoma
  * Leukemic phase (> 5,000 malignant lymphocytes/µl)
  * Mass over 5 cm in greatest diameter
  * For lymphoplasmacytic lymphoma: additional treatment criteria are serum viscosity ≥ 4 cp, serum monoclonal protein > 5 g/L, concurrent primary systemic AL amyloidosis, cold agglutinin disease
* Age over 18
* Prior treatment with bortezomib and/or rituximab is acceptable
* For follicular lymphoma only, at least one prior treatment

Exclusion Criteria:

* Platelet count of < 100 X10 /L within 14 days before enrollment, unless due to bone marrow infiltration with lymphoma, or due to autoimmune thrombocytopenia because of lymphoma.
* Patient has an absolute neutrophil count of < 1.0 X 10/L within 14 days before registration, unless due to bone marrow infiltration with lymphoma.
* Patient has a calculated or measured creatinine clearance of <20 mL/minute within 14 days before registration. (Creatinine Clearance is indicated through the Serum Creatinine. If the Serum Creatinine is abnormal, the physician may then due a 24 hour urine to further clarify Creatinine Clearance. A 24 hour urine test is not required per study.)
* Patient has ≥ Grade 2 peripheral neuropathy within 14 days before registration.
* Myocardial infarction within 6 months prior to registration or has New York Heart Association (NYHA) Class III or IV heart failure. uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant
* Patient received other investigational drugs with 14 days before registration
* Serious medical or psychiatric illness likely to interfere with study participation
* Diagnosed or treated for another malignancy within 3 years of registration, w/ the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* CNS involvement with lymphoma.
* Known HIV-positive.
* History of disease refractory to a purine analog (defined as remission duration of < 6 months to therapy that included fludarabine, pentostatin, or cladribine).
* History of intolerance of bortezomib, boron, mannitol, cladribine, or rituximab.
* Patient has > 1.5 X ULN Total Bilirubin
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07-07 (Actual); Primary Completion 2014-09-12 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O. Persky, MD, Principal Investigator — University of Arizona
Locations (1):
- The University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Puvvada SD, Guillen-Rodriguez J, Kumar A, Inclan L, Heard K, Rivera XI, Anwer F, Schatz JH, Mahadevan D, Persky DO. Phase 2 Open-Label Study of Bortezomib, Cladribine, and Rituximab in Advanced, Newly Diagnosed, and Relapsed/Refractory Mantle-Cell and Indolent Lymphomas. Clin Lymphoma Myeloma Leuk. 2018 Jan;18(1):58-64. doi: 10.1016/j.clml.2017.09.001. Epub 2017 Sep 19. PMID 29056470

RESULTS

PARTICIPANT FLOW:
Groups:
- VCR (Velcade, Cladribine and Rituximab): * Rituximab 375 mg/m2 IV day1
  * Cladribine 4 mg/m2 IV over 2 hours days 1-5
  * Bortezomib 1.3 mg/m2 IV days 1 and 4
  * Repeat every 28 days for a maximum of 6 cycles
  rituximab: 375 mg/m2 IV Day 1. Repeat every 28 days for a maximum of 6 cycles.
  bortezomib: 1.3 mg/m2 IV Days 1 and 4. Repeat every 28 days for a maximum of 6 cycles.
  cladribine: 4 mg/m2 IV over 2 hours Days 1-5. Repeat every 28 days for a maximum of 6 cycles.
Period: Overall Study
Arm/Group | VCR (Velcade, Cladribine and Rituximab)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VCR (Velcade, Cladribine and Rituximab)
Number analyzed (Participants) | 24
Age, Continuous [Median (Standard Deviation); unit: years] | 66.5 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Histology [Count of Participants; unit: Participants]
  Mantle-cell lymphoma | 11
  Follicular lymphoma | 5
  Marginal zone lymphoma | 4
  Lymphoplasmacytic lymphoma | 3
  Small lymphocytic lymphoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 2 Years
Description: PFS was calculated from the first dose of study drug to the first documentation of disease progression, death regardless of cause, or change in therapy due to disease progression, whichever occurred first. If disease progression did not occur by the end of treatment, patients were evaluated every 3 months until progression with physical examination, laboratory studies, and conventional computed tomographic imaging, up to a maximum of 2 years. The Kaplan-Meier product-limit method will be used to estimate progression-free survival in the presence of censoring.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | VCR (Velcade, Cladribine and Rituximab)
Number analyzed (Participants) | 23
Participants | 15

2. Secondary Outcome: Overall Survival at 2 Years
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | VCR (Velcade, Cladribine and Rituximab)
Number analyzed (Participants) | 23
Participants | 18

3. Secondary Outcome: Complete Response Rate
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | VCR (Velcade, Cladribine and Rituximab)
Number analyzed (Participants) | 23
Participants | 8

4. Secondary Outcome: Partial Response
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | VCR (Velcade, Cladribine and Rituximab)
Number analyzed (Participants) | 23
Participants | 14

ADVERSE EVENTS:
Time Frame: 107 months
Arm/Group | VCR (Velcade, Cladribine and Rituximab)
All-Cause Mortality (participants affected / at risk) | 8/24
Serious Adverse Events (participants affected / at risk) | 14/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VCR (Velcade, Cladribine and Rituximab) (N=24)
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 5
Anemia (Blood and lymphatic system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VCR (Velcade, Cladribine and Rituximab) (N=24)
Fatigue (General disorders) | 19
Fever (General disorders) | 4
Neuropathy (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT00980395/Prot_SAP_000.pdf